CLINICAL TRIAL: NCT02313571
Title: Incidence and Characteristics of Breakthrough Pain in Parturients Using Computer Integrated Patient Controlled Epidural Analgesia
Brief Title: Breakthrough Pain Computer Integrated Patient Controlled Epidural Analgesia
Acronym: BTP
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012/061/D
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Epidural Analgesia; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The computer-integrated patient controlled epidural analgesia (CIPCEA) system can automatically adjust the background infusion rate during combined spinal-epidural (CSE) analgesia based on the parturient's need as labour progresses. Analysis of parturients experiencing breakthrough pain may identify associated factors that can also be related to obstetric or foetal outcomes

DETAILED DESCRIPTION:
Computer integrated patient controlled epidural analgesia (CIPCEA) is a novel epidural analgesic delivery system that is currently used in daily practice in KK Women's and Children's Hospital. It has enabled us to monitor the infusion pumps through wireless connection to a central monitoring system and hence, collect pump utilisation data electronically. The CIPCEA system is programmed to analyse the LA usage across the last hour and adjust the background infusion rate according to a preset algorithm.

Breakthrough pain is defined as maternal complaint of pain or pressure that required and was successfully treated with supplemental epidural medications. we investigated the potential factors associated with breakthrough pain in patients who receive CSE epidural analgesia with CIPCEA, with the aim of elucidating the important associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women,
* requested for epidural analgesia

Exclusion Criteria:

* Multiparous women,
* unable to perform combined spinal epidural technique

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who had nulliparous requested for labour epidural analgesia
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2010-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Breakthrough Pain (Requiring unscheduled epidural supplementation by anaesthetists) | 1 day
  Requiring unscheduled epidural supplementation by anaesthetists

SECONDARY OUTCOMES:
Caesarean Section (Rate of caesarean section) | 1 day
  Rate of caesarean section
Instrumental Delivery (Rate of instrumental delivery) | 1 day
  Rate of instrumental delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore